CLINICAL TRIAL: NCT06952946
Title: Effects of Different Fresh Gas Flow Applications on Postoperative Nausea and Vomiting in Septorhinoplasty Surgeries
Brief Title: Effect of Fresh Gas Flow Differences on Postoperative Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Ufuk Karbaş, Specialist physician, Adiyaman University Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AURH-AR-UK-01
Record Dates: First submitted 2025-04-14; First posted 2025-05-01 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Nausea and Vomiting, Postoperative; Septoplasty/Septorhinoplasty
Keywords: fresh gas flow; low flow anesthesia; postoperative nausea vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: Three groups to which fresh gas flow is applied as low flow (0.5 l/min), medium flow (2 l/min) and high flow (4 l/min).
Who Masked: Participant
Masking Description: Researchers who will evaluate postoperative nausea and vomiting and patients participating in the study will be blinded to the difference in fresh gas flow that will be applied to them.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low flow anesthesia group (Active Comparator): After endotracheal intubation, fresh gas flow will be applied at 4 lt/min for 8 minutes, and in the low-flow anesthesia group, it will be reduced to 0.5 lt/min and maintained at this flow throughout the surgery.
  Interventions: Other: 0.5 lt/dk fresh gas flow
- medium flow anesthesia group (Active Comparator): After endotracheal intubation, fresh gas flow will be applied at 4 lt/min for 8 minutes, and in the medium-flow anesthesia group, it will be reduced to 2 lt/min and maintained at this flow throughout the surgery.
  Interventions: Other: 2 lt/dk fresh gas flow
- high flow anesthesia group (Active Comparator): After endotracheal intubation, fresh gas flow will be applied at 4 lt/min for 8 minutes and then continued in the same manner (4 lt/min) in the high-flow anesthesia group.
  Interventions: Other: 4 lt/dk fresh gas flow

INTERVENTIONS:
Other: 0.5 lt/dk fresh gas flow — Fresh gas flow will be set to 0.5 l/min in the low flow anesthesia group.
  Arms: low flow anesthesia group
Other: 2 lt/dk fresh gas flow — Fresh gas flow will be set to 2 lt/min in the medium flow anesthesia group.
  Arms: medium flow anesthesia group
Other: 4 lt/dk fresh gas flow — Fresh gas flow will be set to 4 lt/min in the high flow anesthesia group.
  Arms: high flow anesthesia group

SUMMARY:
The aim of this study is to investigate the effect of fresh gas flow applied during general anesthesia on the incidence of postoperative nausea and vomiting in patients undergoing septorhinoplasty surgery. Patients who agree to participate in the study will be divided into three groups according to the fresh gas flow applied: low flow (0.5 lt/min) (Group L), medium flow (2 lt/min) (Group M) and high flow (4 lt/min) (Group H), and the postoperative nausea and vomiting data of the groups will be compared.

DETAILED DESCRIPTION:
Preoperative demographic characteristics and Apfel score (smoking history, gender, postoperative opioid use, POB history) of the patients will be recorded. General anesthesia will be applied to all patients with standard ASA monitoring. In general anesthesia induction, 2 mg/kg propofol, 1 mcg/kg remifentanil, 0.6 mg/kg rocuronium will be used for all patients. Sevoflurane (minimum alveolar concentration of 1) will be used as a volatile agent and remifentanil (0.1 mcg-1 mcg/kg/h) will be used as an analgesic agent for anesthesia maintenance. After endotracheal intubation, fresh gas flow will be applied at 4 lt/min for 8 minutes, reduced to 0.5 lt/min in Group L, 2 lt/min in Group M, and maintained at 4 lt/min in Group H. After extubation, patients will be monitored in the recovery unit for at least 30 minutes, and at postoperative 0th minute (when first seen in the recovery room), 30th minute, 1st hour, 6th hour, 12th hour and 24th hour, the nausea score of the patients will be evaluated using the Numerical Rating Scale (NRS) with a score between 0 and 10. If vomiting is present, the number of times the patient vomited will be questioned and recorded. The patients' postoperative VAS scores, the amount of antiemetics used, the amount of opioids used intraoperatively and postoperatively will be recorded, and comparisons will be made between the groups and evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agreed to participate in the study
* 18-65 years of age
* ASA I-II risk group patients

Exclusion Criteria:

* Patient does not accept the study
* Presence of psychiatric disorder and patient's inability to cooperate
* Cognitive dysfunction
* Hearing problems
* History of alcohol or drug addiction
* Presence of a serious pre-existing medical condition that limits objective assessment
* Complications developed during surgery
* Presence of any life-threatening condition after surgery
* Patient's classification is ASA III-IV

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-09-28 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
postoperative nausea and vomiting | 24 hours
  The patients' postoperative nausea and vomiting scores will be assessed when they are taken to the postoperative care room, immediately before being transferred from the postoperative care room to the ward (at the 30th minute postoperatively), at the 1st hour postoperatively, at the 6th hour postoperatively, at the 12th hour postoperatively, and at the 24th hour postoperatively. Nausea will be assessed by scoring with a numerical rating scale between 0 and 10. Vomiting will be questioned. If vomiting occurs, the number of times it occurs will be questioned. Whether postoperative antiemetics are used and if so, how many mg are used will be recorded. If postoperative opioids are used, how many mg are used will be recorded.

SECONDARY OUTCOMES:
intraoperative body temperature | intraoperative
  Intraoperative body temperature values of patients in all groups will be monitored throughout the operation with a thermometer probe placed under the right armpit; axillary body temperature will be recorded every 5 minutes in the first half hour, 10 minutes in the next half hour, and every half hour after the first hour. Body temperature changes of the groups will also be compared.
Whether kidney functions are affected | 1 hour postoperative
  By comparing the kidney function tests (urea-creatinine) of the patients before and after the surgery (postoperative 1st hour), it will be evaluated whether the flow differences (especially low flow) have any negative effects on kidney functions.
whether liver functions are affected | 1 hour postoperative
  Patients' liver function tests (AST-ALT) before and after surgery (postoperative 1st hour) will be compared to evaluate whether flow differences (especially low flow) have any negative effects on liver functions.

CONTACTS AND LOCATIONS:
Locations (1):
- Adıyaman Training and Research Hospital, Adıyaman, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No